CLINICAL TRIAL: NCT02063737
Title: The Sleep Track Text Pilot Trial in Emergency Care Clinicians
Brief Title: SleepTrackTXT Feasibility and Pilot Study
Acronym: SleepTrackTXT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Daniel Patterson, PhD, NREMT-P, Assistant Professor of Emergency Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO13120428
Record Dates: First submitted 2014-01-10; First posted 2014-02-14 (Estimated); Results first posted 2015-07-13 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-07

CONDITIONS: Fatigue
Keywords: Shift work; Fatigue; Sleepiness; Injury
MeSH Terms: conditions — Fatigue; Sleepiness; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Sham Comparator): The control group will receive text-message assessments only at the start, during, and end of shift. These queries will attempt to capture the worker's self-reported sleepiness, fatigue, and occurrence of work-related injury during shift work.
  Interventions: Behavioral: Text-message assessments only
- Intervention Group (Experimental): The intervention group will receive the same text-message assessments as the control group. In addition, these subjects will receive text-message interventions for high level fatigue for reducing fatigue and sleepiness during shift work if they report a high-level of fatigue or sleepiness at the start or during their shift. These subjects will then receive additional text message queries at the end of their shifts to determine if they adopted a strategy for reducing perceived sleepiness or fatigue.
  Interventions: Behavioral: Text-message interventions for high level fatigue

INTERVENTIONS:
Behavioral: Text-message assessments only — Text message assessments only. No intervention for high level fatigue.
  Arms: Control Group
Behavioral: Text-message interventions for high level fatigue — Intervention messages to promote alertness while on duty at work including activities. Additionally at the end of the shift, participants were queried on their adoption of the suggested activities and perception of the activities' effectiveness.
  Arms: Intervention Group

SUMMARY:
Aim 1: To determine if real-time assessments of perceived sleepiness and fatigue using text-messaging impacts an emergency medicine clinician's Attitudes, Perceived Norms, Self-Efficacy, Alertness Habits, Perceived Importance of Fatigue, Knowledge of Sleepiness/Fatigue, and Perceptions of Environmental Constraints regarding behaviors that can improve alertness during shift work.

Aim 2: To determine if text-messaging emergency care workers fatigue-reduction strategies in real-time at the start and during shift work reduces worker perceived sleepiness and fatigue at the end of shift work.

DETAILED DESCRIPTION:
More than half (55%) of Emergency Medical Services (EMS) shift workers report severe mental and physical fatigue while at work,(Patterson et al, 2012) 36% report excessive daytime sleepiness,(Pirrallo et al; 2012) and 60% poor sleep quality.(Patterson et al; 2012) Sleepiness or fatigue while on duty can result in injuries to EMS workers and medical errors for patients.(Patterson et al; 2012) The investigators' recent research shows that odds of injury among fatigued EMS workers are 1.9 times higher than non-fatigued workers.(Patterson et al; 2012) Additional data show that other emergency workers (e.g., emergency physicians and nurses) are vulnerable to sleepiness and fatigue while at work.(Fisman et al; 2007; Machi et al; 2012; Thomas et al; 2006; Geiger-Brown et al; 2012).

There are a number of individual and system factors that influence sleepiness and fatigue during shift work for emergency workers. Individual factors include sleep hygiene, medical conditions like obstructive sleep apnea, and other factors.(Schaefer et al; 2012; Simon et al; 2012) System factors include shift length, patient care intensity, and workload. Many factors are modifiable, yet some are more difficult than others to change or control. Reducing shift length and customary patterns of shift work, such as 12-hr and 24-hr shifts, is not feasible for many employers and shift workers in the emergency medicine care setting. In some locations, >80% of EMS workers hold multiple jobs, 40% work more than 16 shifts per month, and many accumulate unsafe amounts of overtime in order to make a livable wage.(Patterson et al, 2010; Patterson et al, 2012; Bauder 2012) Other shift workers in emergency care settings face the same or similar obstacles as do EMS shift workers.

An objective of this research study is to pilot test real-time assessment of emergency care worker sleepiness and fatigue. The investigators seek to determine if text-messaging fatigue-reduction strategies to emergency care workers that report a high-level of sleepiness or fatigue at the start or during their shift reduces perceived sleepiness or fatigue at the end of shift. A long term goal of this research is to determine if this innovative text-messaging tool can be used to reduce the likelihood of fatigue-related injury among emergency care shift workers.

Aim 1: To determine if real-time assessments of perceived sleepiness and fatigue using text-messaging impacts a worker's Attitudes, Perceived Norms, Self-Efficacy, Alertness Habits, Perceived Importance of Fatigue, Knowledge of Sleepiness/Fatigue, and Perceptions of Environmental Constraints regarding behaviors that can improve alertness during shift work.

Rationale: The investigators recognize that emergency care shift workers hold different beliefs and attitudes about the risk of sleepiness and fatigue on duty and are at different stages of adopting risk-reduction behaviors. Behavioral research shows that modifying one or more of these factors can impact future behavior and potentially reduce risk over the long term. Approach: The investigators have developed a list of candidate items that operationalize the Integrative Model of Behavioral Prediction. The investigators will administer these candidate items at baseline and again at the end of the study period to assess impact.

Aim 2: To determine if text-messaging emergency care workers fatigue-reduction strategies in real-time at the start and during shift work reduces worker perceived sleepiness and fatigue at the end of shift work.

Approach: At baseline, the investigators will randomly assign 100 emergency care workers to one of two groups (the control group or intervention group). The control group (n=50 / 50%) will receive standard text-message questions of sleepiness and fatigue at the beginning, during, and end of shift. The other 50% (n=50) will be assigned to our intervention group and receive the same text-message questions as the control group, as well as additional text-messages that include strategies that the investigators hypothesize will lead to a reduction in perceived sleepiness or fatigue at the end of shift work. With 100 EMS workers (50% intervention / 50% control), the investigators have 80% power to detect a difference (effect size of 0.78) in the self-reported fatigue levels reported at the end of shift by the control and intervention groups. The investigators will collect data over a 90-day study period.

Eligibility Criteria include:

1. The study subject must be 18 years of age or older;
2. The study subject must currently work in the emergency medicine setting as an emergency physician, emergency nurse, or emergency medical technician (EMT) / paramedic worker;
3. The study subject must work shifts as part of your employment in the emergency medicine setting;
4. The study subject must have a cell-phone / smartphone that can receive and send text-messages;
5. The study subject must be willing to take part in a research study where he/she is required to send and receive multiple text-messages at the start, during, and end of scheduled shift work?

ELIGIBILITY:
Inclusion Criteria:

1. Are 18 years of age or older;
2. Currently work in the emergency medicine setting as an emergency physician, emergency nurse, or emergency medical technician (EMT) / paramedic worker;
3. Currently working shifts as part of your employment in the emergency medicine setting;
4. Have a cell-phone / smartphone that can receive and send text-messages;
5. Willing to take part in a research study where you are required to send and receive multiple text-messages at the start, during, and end of your shift work?

Exclusion Criteria:

1: Those that do not meet inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Patterson, PhD, Principal Investigator — University of Pittsburgh Department of Emergency Medicine School of Medicine
Locations (1):
- University of Pittsburgh Department of Emergency Medicine School of Medicine, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Patterson PD, Moore CG, Weaver MD, Buysse DJ, Suffoletto BP, Callaway CW, Yealy DM. Mobile phone text messaging intervention to improve alertness and reduce sleepiness and fatigue during shiftwork among emergency medicine clinicians: study protocol for the SleepTrackTXT pilot randomized controlled trial. Trials. 2014 Jun 21;15:244. doi: 10.1186/1745-6215-15-244. PMID 24952387
- [Result] Patterson PD, Buysse DJ, Weaver MD, Callaway CW, Yealy DM. Recovery between Work Shifts among Emergency Medical Services Clinicians. Prehosp Emerg Care. 2015 Jul-Sep;19(3):365-75. doi: 10.3109/10903127.2014.995847. Epub 2015 Feb 6. PMID 25658148
- [Result] Patterson PD, Klapec SE, Weaver MD, Guyette FX, Platt TE, Buysse DJ. Differences in Paramedic Fatigue before and after Changing from a 24-hour to an 8-hour Shift Schedule: A Case Report. Prehosp Emerg Care. 2016;20(1):132-6. doi: 10.3109/10903127.2015.1025158. Epub 2015 May 15. PMID 25978152
- [Result] Patterson PD, Buysse DJ, Weaver MD, Doman JM, Moore CG, Suffoletto BP, McManigle KL, Callaway CW, Yealy DM. Real-time fatigue reduction in emergency care clinicians: The SleepTrackTXT randomized trial. Am J Ind Med. 2015 Oct;58(10):1098-113. doi: 10.1002/ajim.22503. Epub 2015 Aug 25. PMID 26305869
- [Derived] Patterson PD, Moore CG, Guyette FX, Doman JM, Sequeira D, Werman HA, Swanson D, Hostler D, Lynch J, Russo L, Hines L, Swecker K, Runyon MS, Buysse DJ. Fatigue mitigation with SleepTrackTXT2 in air medical emergency care systems: study protocol for a randomized controlled trial. Trials. 2017 Jun 5;18(1):254. doi: 10.1186/s13063-017-1999-z. PMID 28583143

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: The control group will receive text-message queries at the start, during, and end of shift. These queries will attempt to capture the worker's self-reported sleepiness, fatigue, and occurrence of work-related injury during shift work.
- Intervention Group: The intervention group will receive the same text-message queries as the control group. In addition, these subjects will receive suggestions (strategies) for reducing fatigue and sleepiness during shift work if they report a high-level of fatigue or sleepiness at the start or during their shift. These subjects will then receive additional text-message queries at the end of their shifts to determine if they adopted a strategy for reducing perceived sleepiness or fatigue.
  Text-message strategies: If an intervention subject reports a high level of sleepiness or fatigue at the start or during their shift work, these subjects will receive additional text-messages that include strategies (suggestions) for reducing perceived fatigue or sleepiness during shift work. These subjects will also receive an additional text-message at the end of their shift to determine if the subject adopted the strategy suggested and if it helped reduced perceived fatigue or sleepiness.
Period: Overall Study
Arm/Group | Control Group | Intervention Group
Started | 52 | 48
Completed | 41 | 44
Not Completed | 11 | 4
Not completed — Lost to Follow-up | 11 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention Group | Total
Number analyzed (Participants) | 52 | 48 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (10.2) | 35.0 (9.7) | 35.6 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 18 | 29
  Male | 41 | 30 | 71
Certification/License [Number; unit: participants]
  EMT-Basic | 4 | 5 | 9
  Paramedic | 34 | 31 | 65
  Nurse | 7 | 10 | 17
  Physician/Other | 7 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Self-Reported Fatigue at End of Shift Work
Description: Self-reported fatigue based on scale ranging from 0 (Not At All) to 5 (Very Much).
Time Frame: At the end of scheduled work shifts during a 90 day study period
Population: Analysis using intention to treat.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Units Other Than Participants: Shifts
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 51 | 47
Number analyzed (Shifts) | 1389 | 1232
units on a scale | 2.17 (0.1746) | 1.78 (0.1782)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Superiority or Other; p = 0.0830, Mixed Models Analysis; adjusting for shift length; Median Difference (Final Values) = -0.3882, 95% CI 2-sided [-0.8272 to 0.0508] — Adjusted difference between intervention groups (intervention - control) from the linear mixed model adjusting for shift length and repeated measures within individuals

2. Secondary Outcome: Attitude One Subscale of the Sleep Fatigue and Alertness Behavior (SFAB) Tool
Description: Individual attitudes towards maintaining alertness and reducing fatigue at work. Scale ranges from 0 to 100 with higher scores indicating a more positive/favorable attitude towards maintaining alertness and reducing fatigue while at work.
Time Frame: Assessed at the end of 90-day study period
Population: Intention to treat among participants with 90 day data (completers)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 41 | 44
units on a scale | 61.9 (19.9) | 69.3 (17.1)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Superiority or Other; p = 0.0114, ANCOVA; adjusting for baseline measure

3. Secondary Outcome: Attitudes Two Subscale of the Sleep Fatigue and Alertness Behavior Tool
Description: Individual attitudes towards maintaining alertness and reducing fatigue at work on future shifts. Scale ranges from 0 to 100 with higher scores indicating a more positive/favorable attitude towards maintaining alertness and reducing fatigue while at work.
Time Frame: end of study at 90 day follow up
Population: Intention to treat among participants with 90 day data (completers)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 41 | 44
units on a scale | 27.8 (21.1) | 30.3 (22.8)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Superiority or Other; p = .99, ANCOVA; adjusting for the baseline measure

4. Secondary Outcome: Normative Beliefs Scale One Subscale of the SFAB
Description: Belief of people's views if they thought you were sleepy and fighting the urge to sleep while at work. Scale ranges from 0 (strongly approve) to 100 (strongly disapprove). Higher scores indicate a person believes the social norms and beliefs of his/her social network possess a negative view of behaviors that places an individual at work while very sleepy or fatigued.
Time Frame: end of study at 90 day follow up
Population: Intention to treat among participants with 90 day data (completers)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 41 | 44
units on a scale | 48.9 (18.8) | 59.7 (18.8)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Superiority or Other; p = 0.0927, ANCOVA; adjusted for baseline measure

5. Secondary Outcome: Normative Beliefs Scale Two Subscale of the SFAB
Description: Belief of people's views if they thought you were very fatigued mentally or physically while at work. Scale ranges from 0 (strongly approve) to 100 (strongly disapprove). Higher scores indicate a person believes the social norms and beliefs of his/her social network possess a negative view of behaviors that places an individual at work while very sleepy or fatigued.
Time Frame: end of study at 90 day follow up
Population: Intention to treat among participants with 90 day data (completers)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 41 | 44
units on a scale | 47.2 (19.8) | 58.8 (25.6)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Superiority or Other; p = 0.0578, ANCOVA; adjusting for the baseline measure

6. Secondary Outcome: Self Efficacy Subscale of the SFAB
Description: Degree of confidence from 0 (cannot do at all) to 100 (highly certain can do) for completing activities. Higher scores indicate the individual has a high-level of self-confidence he/she can perform select behaviors that may improve alertness and reduce feelings of sleepiness or fatigue while at work.
Time Frame: end of study at 90 day follow up
Population: Intention to treat among participants with 90 day data (completers)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 41 | 44
units on a scale | 57.9 (24.9) | 58.9 (26.8)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Superiority or Other; p = 0.69, ANCOVA; adjusting for baseline measure

7. Secondary Outcome: Knowledge-one Subscale of SFAB
Description: Perception that fatigue and sleepiness at work increases risks to safety ranging from 0 (strongly disagree) to 100 (strongly agree). Higher scores indicate an individual has a high-level of awareness for the negative effects of sleepiness and fatigue while at work, that may be attributed to the acquisition of information, an increased understanding, or through experiences or education.
Time Frame: end of study at 90 day follow up
Population: Intention to treat among participants with 90 day data (completers)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 41 | 44
units on a scale | 76.5 (22.5) | 81.4 (19.5)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Superiority or Other; p = 0.65, ANCOVA; adjusting for baseline measure

8. Secondary Outcome: Knowledge-two Subscale of the SFAB
Description: Perceived degree of evidence that fatigue and sleepiness at work increases risks to safety ranging from 0 (strongly disagree) to 100 (strongly agree). Higher scores indicate an individual has a high-level of awareness for the negative effects of sleepiness and fatigue while at work, that may be attributed to the acquisition of information, an increased understanding, or through experiences or education.
Time Frame: end of study at 90 day follow up
Population: Intention to treat among participants with 90 day data (completers)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 41 | 44
units on a scale | 77.1 (17.8) | 76.8 (18.3)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Superiority or Other; p = 0.95, ANCOVA; adjusting for baseline measure

9. Secondary Outcome: Importance Subscale of SFAB
Description: Level of importance an individual places on the need to maintain alertness and reduce feelings of fatigue and/or sleepiness while at work ranging from 0 (strongly disagree) to 100 (strongly agree). Strongly agree (higher score) is associated with high level of importance (endorsement) placed on the need to maintain alertness and reduce feelings of fatigue while at work.
Time Frame: end of study at 90 day follow up
Population: Intention to treat among participants with 90 day data (completers)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 41 | 44
units on a scale | 62.0 (16.5) | 68.8 (18.6)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Superiority or Other; p = 0.21, ANCOVA; adjusting for baseline measure

10. Secondary Outcome: Environmental Constraints One Subscale of the SFAB
Description: Degree of importance of employer based barriers that might limit ability to reduce feelings of fatigue and sleepiness while on duty. Scale ranges from 0 (not at all important) to 100 (very important). Higher scores indicate the individual perceives his/her employer's policies and organizational related procedures/protocols as factors that inhibit the individual's ability to engage in behaviors that can improve alertness and reduce feelings of sleepiness or fatigue while at work.
Time Frame: end of study at 90 day follow up
Population: Intention to treat among participants with 90 day data (completers)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 41 | 44
units on a scale | 64.5 (27.5) | 64.4 (29.6)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Superiority or Other; p = 0.51, ANCOVA; adjusting for baseline measure

11. Secondary Outcome: Environmental Constraints Two Subscale of the SFAB
Description: Degree of importance of employer policies that might limit ability to reduce feelings of fatigue and sleepiness while on duty. Scale ranges from 0 (not at all important) to 100 (very important). Higher scores indicate the individual perceives his/her employer's policies and organizational related procedures/protocols as factors that inhibit the individual's ability to engage in behaviors that can improve alertness and reduce feelings of sleepiness or fatigue while at work.
Time Frame: end of study at 90 day follow up
Population: Intention to treat among participants with 90 day data (completers)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 41 | 44
units on a scale | 38.3 (31.1) | 45.5 (33.4)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Superiority or Other; p = 0.28, ANCOVA; adjusting for baseline measure

12. Secondary Outcome: Environmental Constraints Three Subscale of the SFAB
Description: Degree of importance of personal/work-life barriers that might limit ability to reduce feelings of fatigue and sleepiness while on duty. Scale ranges from 0 (not at all important) to 100 (very important). Higher scores indicate the individual perceives his/her responsibilities unrelated to the organization as factors that inhibit the individual's ability to engage in behaviors that can improve alertness and reduce feelings of sleepiness or fatigue while at work
Time Frame: end of study at 90 day follow up
Population: Intention to treat among participants with 90 day data (completers)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 41 | 44
units on a scale | 49.4 (24.4) | 44.5 (23.0)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Superiority or Other; p = 0.0930, ANCOVA; adjusting for baseline measure

13. Secondary Outcome: Habits Subscale of the SFAB
Description: Endorsement of behaviors that may promote improved alertness and reduced feelings of sleepiness or fatigue while at work ranging from 0 (strongly agree) to 100 (strongly disagree). Strongly agree (lower score) is associated with high level of endorsement of behaviors (habits) that promote improved alertness.
Time Frame: end of study at the 90 day follow up
Population: Intention to treat among participants with 90 day data (completers)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 41 | 44
units on a scale | 39.3 (21.6) | 48.5 (26.8)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Superiority or Other; p = 0.56, ANCOVA; adjusting for baseline measure

14. Secondary Outcome: Intentions Subscale of the SFAB
Description: An individual's intent to engage in behaviors that may promote improved alertness and reduced feelings of sleepiness or fatigue while at work with higher scores indicating greater intent. Range is 0 (strongly agree) to 100 (strongly disagree).
Time Frame: end of study at 90 day follow up
Population: Intention to treat among participants with 90 day data (completers)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 41 | 44
units on a scale | 72.3 (14.7) | 77.4 (17.0)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Superiority or Other; p = 0.20, ANCOVA; adjusting for baseline measure

ADVERSE EVENTS:
Arm/Group | Control Group | Intervention Group
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/48
Other Adverse Events (participants affected / at risk) | 0/52 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No